CLINICAL TRIAL: NCT05478694
Title: Prospective Single Institutional Study Evaluating the Outcomes for Patients Undergoing Ablative Therapies in the Management of Clinically Localized Prostate Cancer in the Primary and Salvage Setting
Brief Title: Outcomes of Focal Ablation for Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Xiaosong Meng, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2022-0641
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Focal ablation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: US Export: No

GROUPS / COHORTS (1):
- Ablative Therapy Group: Enrolled subjects will undergo the ablative therapy as part of their standard of care treatment

SUMMARY:
This study will be designed to define the efficacy and safety of ablative therapies in the management of localized prostate cancer and comprehensively evaluate quality of life outcomes and oncologic control following treatment.

DETAILED DESCRIPTION:
This study will be designed to define the efficacy and safety of ablative therapies in the management of localized prostate cancer and comprehensively evaluate quality of life outcomes and oncologic control following treatment.

There are several commercially available standard of care treatments available for local therapy of the prostate. Ablative therapies may be delivered via a whole gland or focal approach by systems including cryoablation (CA), brachytherapy, irreversible electroporation (IRE), high intensity focused ultrasound (HIFU), MRI-guided transurethral ultrasound ablation (TULSA) procedure or future novel prostate ablation systems.

These are single, outpatient treatments lasting between 2-4 hours and include treatment planning and energy delivery under guidance and are either administered via transperineally approach (cryoablation, IRE, brachytherapy) or via the urethral (TULSA-Pro) or rectum (HIFU).

This study protocol will not include experimental therapy and the enrolled subjects will undergo the ablative therapy as part of their standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men with histologically confirmed prostate adenocarcinoma diagnosed on prostate biopsy
* Men with histologically confirmed local recurrence of prostate cancer diagnosed on prostate biopsy and standard of care imaging excluding locoregional or metastatic disease
* Age 18-90 years.
* Life expectancy > 1 year
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Anatomic abnormalities that do not allow for focal ablation
* Evidence of non-organ confined disease that is not feasible for ablation
* Has active urinary traction infection

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Oncologic outcomes as assessed by the rate of negative in-field biopsy at 12 months (primary setting) | 12 months post treatment
  Oncologic outcomes will be assessed by the rate of negative in-field biopsy at 12 months which is defined by the Delphi consensus criterion of absence of clinically significant disease (≤ 3 mm of Gleason ≤ 6 disease in any biopsy core is insignificant)
Oncologic outcomes as assessed by the rate of advancement to systemic therapy or radical salvage therapies (primary setting) | 3 years post treatment
  Oncologic outcomes will be assessed by the rate of advancement to systemic therapy or radical salvage therapies which is defined by prostatectomy, radiation or hormone therapy.
Oncologic outcomes as assessed by the rate of negative in-field biopsy at 12 months (salvage setting) | 12 months post treatment
  Oncologic outcomes will be assessed by the rate of negative in-field biopsy at 12 months which is defined by the Delphi consensus criterion of absence of clinically significant disease (≤ 3 mm of Gleason ≤ 6 disease in any biopsy core is insignificant)
Oncologic outcomes as assessed by the rate of progression to systemic therapy or radical salvage therapies (salvage setting) | 3 years post treatment
  Oncologic outcomes will be assessed by the rate of progression to systemic therapy or radical salvage therapies which is defined by prostatectomy, radiation or hormone therapy.
Change in urinary function as measured by International Prostate Symptom Score (IPSS) questionnaire (primary setting) | Baseline and 12 months post treatment
  Change in urinary function is measured by International Prostate Symptom Score (IPSS) questionnaire which measures urinary symptoms and continence and the scores range from 0 to 35. A change > 3 points between baseline and follow-up assessments is defined as meaningful for the IPSS. Therefore, increases in IPSS scores larger than 3 points will be categorized as reduced urinary function (worse outcome).
Change in urinary function as measured by International Prostate Symptom Score (IPSS) questionnaire (salvage setting) | Baseline and 12 months post treatment
  Change in urinary function is measured by International Prostate Symptom Score (IPSS) questionnaire which measures urinary symptoms and continence and the scores range from 0 to 35. A change > 3 points between baseline and follow-up assessments is defined as meaningful for the IPSS. Therefore, increases in IPSS scores larger than 3 points will be categorized as reduced urinary function (worse outcome).
Change in erectile function as measured by International Index of Erectile Function (IIEF-5) score questionnaire (primary setting) | Baseline and 12 months post treatment
  Change in erectile function is measured by International Index of Erectile Function (IIEF-5) score questionnaire which classifies patients into five severity levels ranging from none (22-25 points) to severe (5-7 points). Patients whose IIEF-5 levels worsen from baseline to follow-up will be categorized as having reduced erectile function.
Change in erectile function as measured by International Index of Erectile Function (IIEF-5) score questionnaire (salvage setting) | Baseline and 12 months post treatment
  Change in erectile function is measured by International Index of Erectile Function (IIEF-5) score questionnaire which classifies patients into five severity levels ranging from none (22-25 points) to severe (5-7 points). Patients whose IIEF-5 levels worsen from baseline to follow-up will be categorized as having reduced erectile function.

SECONDARY OUTCOMES:
Number of participants with adverse events or short-term complications (primary setting) | 30 days post treatment
  Adverse events (AE)s will be monitored and evaluated by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for 30 days post-treatment
Number of participants undergoing combined treatment of the transitional zone (TZ ) due to bladder outlet obstruction caused by Benign prostatic hyperplasia (BPH) | Baseline and 12 months post treatment
  Number of participants undergoing combined treatment of the transitional zone (TZ ) due to bladder outlet obstruction caused by BPH will be evaluated to determine efficacy of treatment of the transitional zone in patients with lower urinary tract symptoms (LUTS) due to BPH via International Prostate Symptom Score (IPSS) questionnaire
Number of participants with adverse events or short-term complications (salvage setting) | 30 days post treatment
  Adverse events (AE)s will be monitored and evaluated by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for 30 days post-treatment
Number of participants with adverse events or long-term complications (primary setting) | 3 years post-treatment
  An adverse event (AE) will be monitored and evaluated by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for up to 3 years post-treatment
Number of participants with adverse events or long-term complications (salvage setting) | 3 years post-treatment
  An adverse event (AE) will be monitored and evaluated by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for up to 3 years post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaosong Meng, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UTSW, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will plan on sharing patient demographics, treatment modality, treatment oncologic outcomes, post-treatment questionnaire data and adverse events. Specific patient identifiers will be removed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.